CLINICAL TRIAL: NCT05927363
Title: Impact on the Physical Activity Level of Coronary Patients in Phase 3 of a Therapeutic Educational Consolidation Program Involving a "Patient Partner" Associated With a Healthcare Professional. A Randomized Controlled Trial.
Brief Title: Impact on Physical Activity of Coronary Patients in Phase 3 of a Therapeutic Consolidation Educational Program Involving a "Patient Partner" Associated With a Healthcare Professional.
Acronym: P-HEARTNER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APIRES-NIMAO/2022/VV-01
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction
Keywords: Cardiovascular Rehabilitation; Motivation; Physical Activity
MeSH Terms: conditions — Myocardial Infarction; Motor Activity | interventions — Walk Test

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know whether they have been randomized to the group receiving the usual, standard rehabilitation or the group following the Therapeutic Consolidation Educational Program Involving a "Patient Partner" Associated With a Healthcare Professional.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (No Intervention): Patients in Phase 3 of cardiac rehabilitation, undergoing the usual care provided.
- Experimental Group (Experimental): Patients in Phase 3 of cardiovascular rehabilitation, following a therapeutic educational program for consolidation ("patient partner" and a caregiver) as well as the usual care provided.
  Interventions: Other: Therapeutic educational consolidation program in Phase 3 of cardiac rehabilitation associating a patient & caregiver partnership; Other: Teleconsultation at 2 months; Other: Teleconsultation at 4 months; Other: Remote group education workshop; Other: Administration of self-questionnaires: IPAQ, EMAPS, the Exercise Confidence Survey, EQ-5D-5L and the Mediterranean diet adherence score.; Diagnostic Test: 6-minute walk test and administers the modified Borg scale at its conclusion.; Diagnostic Test: Biological check-up; Device: Accelerometer; Other: Administration of a logbook

INTERVENTIONS:
Other: Therapeutic educational consolidation program in Phase 3 of cardiac rehabilitation associating a patient & caregiver partnership — In the experimental group, patients benefit from the usual management as part of the phase 2 post-CR follow-up, with the provision of an information booklet on the benefits of physical activity, and a telephone contact in the event of any questions. In addition, they benefit from the "Consolidation therapeutic education program in phase 3 of CR associating a patient & caregiver partnership, which consists of two teleconsultation sessions at 2 and 4 months, followed by a remote group education workshop co-facilitated by the patient and caregiver partnership at 5 months.
  Discussions during teleconsultations will be recorded to identify the main barriers to physical activity mentioned by patients, and the responses provided by the healthcare professional-peer helper pair during the therapeutic education sessions.
  Arms: Experimental Group
Other: Teleconsultation at 2 months — Discussions during teleconsultations will be recorded to identify the main barriers to physical activity mentioned by patients, and the responses provided by the healthcare professional-peer helper pair during the therapeutic education sessions.
  Arms: Experimental Group
Other: Teleconsultation at 4 months — Discussions during teleconsultations will be recorded to identify the main barriers to physical activity mentioned by patients, and the responses provided by the healthcare professional-peer helper pair during the therapeutic education sessions.
  Arms: Experimental Group
Other: Remote group education workshop — This remote workshop will be co-facilitated by the patient and caregiver partnership at 5 months
  Arms: Experimental Group
Other: Administration of self-questionnaires: IPAQ, EMAPS, the Exercise Confidence Survey, EQ-5D-5L and the Mediterranean diet adherence score. — Patients are then randomly assigned to either the control group (usual management) or the experimental group (management with Patient and Caregiver partnership).
  Arms: Experimental Group
Diagnostic Test: 6-minute walk test and administers the modified Borg scale at its conclusion. — What is a modified Borg scale? The Modified Borg Dyspnea Scale is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administered following a six-minute walking test, one of the most common and frequently used measures to assess disease severity in patients with pulmonary arterial hypertension. Upon conclusion of the 6-minute walking test, the modified Borg scale will be recorded.
  Arms: Experimental Group
Diagnostic Test: Biological check-up — This check-up includes total cholesterol, LDL, HDL, triglycerides, HbA1c.
  Arms: Experimental Group
Device: Accelerometer — An accelerometer is given to the patient, with instructions to wear it for 7 days following the visit (it will then be returned by post).Pre-stamped "bubble" envelopes are given to the patient to return their accelerometer to the measurement points specified in the follow-up.
  Arms: Experimental Group
Other: Administration of a logbook — The patient is given a logbook for daily monitoring of non-measurable physical activities, treatments and medical procedures carried out, as well as any intercurrent events.
  Arms: Experimental Group

SUMMARY:
Following myocardial infarction, cardiac rehabilitation has undeniable benefits on criteria such as cardiovascular mortality and coronary recurrence. Cardiac rehabilitation consists of 3 phases:

1. immediate post-acute, in a cardiology department,
2. active cardiac rehabilitation for several weeks under medical supervision as an inpatient or outpatient,
3. Resumption of active life by the patient. Indeed, one of the major aims of secondary prevention is long-term adherence to physical activity.However, only 20% to 40% of coronary patients remain physically active at 6 months or 1 year, and the effects of Phase 2 cardiac rehabilitation are not maintained. Managing to maintain at least a moderate level of physical activity after Phase 2 of CR is a major objective.

Various interventions (booklets, applications, activity programs, motivational talks led by healthcare professionals have been tested and compared with the usual care in Phase 3 cardiac rehabilitation. An effect seems to exist on the level of physical activity reported, but with a significant evaluation bias. This study aims to use accelerometry to evaluate the 6-month efficacy of the therapeutic education program for consolidation in phase 3 of Cardiovascular Rehabilitation involving a patient partner and a caregiver on moderate-to-sustained physical activity (> 3 METs) in coronary patients on Phase 3 of cardiac rehabilitation compared with usual rehabilitation management.

DETAILED DESCRIPTION:
Following myocardial infarction, cardiac rehabilitation has shown undeniable benefits on strong criteria such as cardiovascular mortality and coronary recurrence. Cardiac rehabilitation consists of 3 phases:

1. immediate post-acute, in a cardiology department,
2. active cardiac rehabilitation for several weeks under medical supervision as an inpatient or outpatient,
3. Resumption of active life by the patient: one of the major aims of secondary prevention is long-term adherence to physical activity.

The importance of phase 2 of cardiac rehabilitation is particularly emphasized and is the subject of recommendations by learned societies. The aim is to re-train the patient under paramedical and medical supervision, and to induce behavioral changes through specific therapeutic education. Exercise re-training aims to increase the patient's cardiorespiratory functional capacity and their ability to do physical activity of moderate-to-sustained intensity. One of the most commonly used units to calculate the intensity of physical activity is the Metabolic Equivalent of Task (MET). The higher the intensity of the activity, the higher the number of METs. Physical activity of at least moderate intensity, as recommended in the long-term care of coronary patients corresponds to 3 METs. The therapeutic objective by international recommendations, and explained to patients during phase 2 CR, is to achieve 150 minutes a week of moderate-to-sustained physical activity (3 METs or more). However, only 20% to 40% of coronary patients remain physically active at 6 months or 1 year, which means that the effects of Phase 2 cardiac rehabilitation are not maintained. Managing to maintain at least a moderate level of physical activity after phase 2 of CR, is a major objective.

Various interventions (booklets, applications, activity programs, motivational talks led by healthcare professionals have been tested and compared with the usual care in Phase 3 cardiac rehabilitation. An effect seems to exist on the level of physical activity reported, but with a significant evaluation bias. Objective, validated measures of physical activity such as accelerometry have not proved their long-term efficacy (6 months being the classically explored endpoint). An intervention establishing a patient-centered relationship and cognitive-behavioral elements would seem to be a perspective of choice to be explored, therapeutic education having been little explored in phase 3 of cardiac rehabilitation and in the long term. To address some of the barriers identified in qualitative studies, the joint participation of a "patient partner" would seem to of interest. The PP is a patient who has acquired knowledge of their disease over time, through experience and experience and therapeutic education. They encourage dialogue between care teams and patients, facilitating patients' self-expression, and contributes to a better understanding of the discourse.

The hypothesis is that a therapeutic educational consolidation program, involving a "patient partner" associated with a health professional, will increase the level of physical activity of coronary patients in Phase 3 of cardiac rehabilitation.

The main objective of this study is to use accelerometry to evaluate the 6-month efficacy of the therapeutic education program for consolidation in phase 3 of Cardiovascular Rehabilitation involving a patient partner and a caregiver on the level of moderate to sustained physical activity (> 3 METs) in coronary patients on Phase 3 of cardiac rehabilitation compared with usual rehabilitation management.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (≥ 18 years).
* Patient having undergone phase 2 treatment in the cardiovascular rehabilitation department of the CHU for myocardial infarction.
* Patient with a means of communication that allows easy internet connection (i.e. a smartphone).
* Patient fluent in French.
* Patient who has given free informed consent.
* Patient affiliated or beneficiary of a health insurance scheme.

Exclusion Criteria:

* Patient with severe or unstable comorbidity (respiratory insufficiency renal failure, decompensated heart failure). heart failure).
* Patient with unstable angina.
* Patient with contraindications to physical activity following physical activity following cardiovascular rehabilitation (according to medical discussion, based on the recommendations of the French Society of Cardiology).
* Patient with no suitable means of communication.
* Patient under court protection, guardianship or curatorship.
* Pregnant, parturient or breast-feeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Moderate-to-sustained physical activity in the Experimental Group | Month 6
  The accelerometer will be used to evaluate the 6-month efficacy of the therapeutic educational program for consolidation in Phase 3 of Cardiovascular Rehabilitation involving a patient partner and a caregiver and its affect on the level of moderate-to-sustained physical activity (> 3 METs) in coronary patients in Phase 3 of cardiac rehabilitation compared with usual rehabilitation management.
  The amount of moderate-to-sustained physical activity (> 3 METs) will be measured in minutes per week.
Moderate-to-sustained physical activity in Controls | Month 6
  The accelerometer will be used to evaluate the 6-month efficacy of the therapeutic educational program for consolidation in Phase 3 of Cardiovascular Rehabilitation involving a patient partner and a caregiver and its affect on the level of moderate-to-sustained physical activity (> 3 METs) in coronary patients in Phase 3 of cardiac rehabilitation compared with usual rehabilitation management.
  The amount of moderate-to-sustained physical activity (> 3 METs) will be measured in minutes per week.

SECONDARY OUTCOMES:
Moderate-to-sustained physical activity in the Experimental Group | Month 3
  The amount of moderate-to-sustained physical activity (> 3 METs) will be measured with the accelerometer in minutes per week.
Moderate-to-sustained physical activity in Controls | Month 3
  The amount of moderate-to-sustained physical activity (> 3 METs) will be measured with the accelerometer in minutes per week.
Number of steps taken per week in the Experimental Group | Month 0
  Number of steps taken per week recorded by the accelerometer
Number of steps taken per week in the Experimental Group | Month 3
  Number of steps taken per week recorded by the accelerometer
Number of steps taken per week in the Experimental Group | Month 6
  Number of steps taken per week recorded by the accelerometer
Number of steps taken per week in Controls | Month 0
  Number of steps taken per week recorded by the accelerometer
Number of steps taken per week in Controls | Month 3
  Number of steps taken per week recorded by the accelerometer
Number of steps taken per week in Controls | Month 6
  Number of steps taken per week recorded by the accelerometer
Time spent sitting/lying down per week in the Experimental Group | Month 0
  Time spent sitting/lying down per week recorded by the accelerometer
Time spent sitting/lying down per week in the Experimental Group | Month 3
  Time spent sitting/lying down per week recorded by the accelerometer
Time spent sitting/lying down per week in the Experimental Group | Month 6
  Time spent sitting/lying down per week recorded by the accelerometer
Time spent sitting/lying down per week in Controls | Month 0
  Time spent sitting/lying down per week recorded by the accelerometer
Time spent sitting/lying down per week in Controls | Month 3
  Time spent sitting/lying down per week recorded by the accelerometer
Time spent sitting/lying down per week in Controls | Month 6
  Time spent sitting/lying down per week recorded by the accelerometer
International Physical Activity Questionnaire Score in the Experimental Group | Month 0
  The short form of the International Physical Activity Questionnaire measures physical activity over the previous week and assesses the types of intensity of physical activity, and sitting time to estimate total physical activity in MET-min/week and time spent sitting. For each category of activity a maximum of 21 hours of activity are permitted a week (3 hours X 7 days).To calculate MET-minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) is multiplied by the number of minutes the activity was carried out, and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET-minutes for that activity are 3.3 X 30 X 5=495 MET-minutes a week. The MET minutes achieved in each category (walking, moderate activity and vigorous activity) are then added together to get the total MET-minutes of physical activity per week.
International Physical Activity Questionnaire Score in the Experimental Group | Month 3
  The short form of the International Physical Activity Questionnaire measures physical activity over the previous week and assesses the types of intensity of physical activity, and sitting time to estimate total physical activity in MET-min/week and time spent sitting. For each category of activity a maximum of 21 hours of activity are permitted a week (3 hours X 7 days).To calculate MET-minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) is multiplied by the number of minutes the activity was carried out, and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET-minutes for that activity are 3.3 X 30 X 5=495 MET-minutes a week. The MET minutes achieved in each category (walking, moderate activity and vigorous activity) are then added together to get the total MET-minutes of physical activity per week.
International Physical Activity Questionnaire Score in the Experimental Group | Month 6
  The short form of the International Physical Activity Questionnaire measures physical activity over the previous week and assesses the types of intensity of physical activity, and sitting time to estimate total physical activity in MET-min/week and time spent sitting. For each category of activity a maximum of 21 hours of activity are permitted a week (3 hours X 7 days).To calculate MET-minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) is multiplied by the number of minutes the activity was carried out, and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET-minutes for that activity are 3.3 X 30 X 5=495 MET-minutes a week. The MET minutes achieved in each category (walking, moderate activity and vigorous activity) are then added together to get the total MET-minutes of physical activity per week.
International Physical Activity Questionnaire Score in Controls | Month 0
  The short form of the International Physical Activity Questionnaire measures physical activity over the previous week and assesses the types of intensity of physical activity, and sitting time to estimate total physical activity in MET-min/week and time spent sitting. For each category of activity a maximum of 21 hours of activity are permitted a week (3 hours X 7 days).To calculate MET-minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) is multiplied by the number of minutes the activity was carried out, and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET-minutes for that activity are 3.3 X 30 X 5=495 MET-minutes a week. The MET minutes achieved in each category (walking, moderate activity and vigorous activity) are then added together to get the total MET-minutes of physical activity per week.
International Physical Activity Questionnaire Score in Controls | Month 3
  The short form of the International Physical Activity Questionnaire measures physical activity over the previous week and assesses the types of intensity of physical activity, and sitting time to estimate total physical activity in MET-min/week and time spent sitting. For each category of activity a maximum of 21 hours of activity are permitted a week (3 hours X 7 days).To calculate MET-minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) is multiplied by the number of minutes the activity was carried out, and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET-minutes for that activity are 3.3 X 30 X 5=495 MET-minutes a week. The MET minutes achieved in each category (walking, moderate activity and vigorous activity) are then added together to get the total MET-minutes of physical activity per week.
International Physical Activity Questionnaire Score in Controls | Month 6
  The short form of the International Physical Activity Questionnaire measures physical activity over the previous week and assesses the types of intensity of physical activity, and sitting time to estimate total physical activity in MET-min/week and time spent sitting. For each category of activity a maximum of 21 hours of activity are permitted a week (3 hours X 7 days).To calculate MET-minutes a week the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) is multiplied by the number of minutes the activity was carried out, and again by the number of days that that activity was undertaken. For example if someone reports walking for 30 minutes 5 days a week then the total MET-minutes for that activity are 3.3 X 30 X 5=495 MET-minutes a week. The MET minutes achieved in each category (walking, moderate activity and vigorous activity) are then added together to get the total MET-minutes of physical activity per week.
Blood pressure in the Experimental Group | Month 0
  mm Hg
Blood pressure in the Experimental Group | Month 3
  mm Hg
Blood pressure in the Experimental Group | Month 6
  mm Hg
Blood pressure in Controls | Month 0
  mm Hg
Blood pressure in Controls | Month 3
  mm Hg
Blood pressure in Controls | Month 6
  mm Hg
Modified Borg score in the Experimental Group | Month 0
  The modified Borg dyspnea score uses a scale from 0 to 10 in which 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6-minute walking test and reflect the maximum degree of dyspnea at any time during the walk test.
Modified Borg score in the Experimental Group | Month 3
  The modified Borg dyspnea score uses a scale from 0 to 10 in which 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6-minute walking test and reflect the maximum degree of dyspnea at any time during the walk test.
Modified Borg score in the Experimental Group | Month 6
  The modified Borg dyspnea score uses a scale from 0 to 10 in which 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6-minute walking test and reflect the maximum degree of dyspnea at any time during the walk test.
Modified Borg score in Controls | Month 0
  The modified Borg dyspnea score uses a scale from 0 to 10 in which 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6-minute walking test and reflect the maximum degree of dyspnea at any time during the walk test.
Modified Borg score in Controls | Month 3
  The modified Borg dyspnea score uses a scale from 0 to 10 in which 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6-minute walking test and reflect the maximum degree of dyspnea at any time during the walk test.
Modified Borg score in Controls | Month 6
  The modified Borg dyspnea score uses a scale from 0 to 10 in which 0 represents no dyspnea and 10 represents maximal dyspnea. Scores are obtained at the end of the 6-minute walking test and reflect the maximum degree of dyspnea at any time during the walk test.
Abdominal circumference in the Experimental Group | Month 0
  In cm
Abdominal circumference in the Experimental Group | Month 3
  In cm
Abdominal circumference in the Experimental Group | Month 6
  In cm
Abdominal circumference in Controls | Month 0
  In cm
Abdominal circumference in Controls | Month 3
  In cm
Abdominal circumference in Controls | Month 6
  In cm
Aerobic capacity in the Experimental Group | Month 0
  Aerobic capacity clinically measured by the 6-minute walking test (number of metres covered).
Aerobic capacity in the Experimental Group | Month 3
  Aerobic capacity clinically measured by the 6-minute walking test (number of metres covered).
Aerobic capacity in the Experimental Group | Month 6
  Aerobic capacity clinically measured by the 6-minute walking test (number of metres covered).
Aerobic capacity in Controls | Month 0
  Aerobic capacity clinically measured by the 6-minute walking test (number of metres covered).
Aerobic capacity in Controls | Month 3
  Aerobic capacity clinically measured by the 6-minute walking test (number of metres covered).
Aerobic capacity in Controls | Month 6
  Aerobic capacity clinically measured by the 6-minute walking test (number of metres covered).
Cholesterol in the Experimental Group | Month 0
  mg/dL
Cholesterol in the Experimental Group | Month 3
  mg/dL
Cholesterol in the Experimental Group | Month 6
  mg/dL
Cholesterol in Controls | Month 0
  mg/dL
Cholesterol in Controls | Month 3
  mg/dL
Cholesterol in Controls | Month 6
  mg/dL
Low-density lipoprotein in the Experimental Group | Month 0
  mg/dL
Low-density lipoprotein in the Experimental Group | Month 3
  mg/dL
Low-density lipoprotein in the Experimental Group | Month 6
  mg/dL
Low-density lipoprotein in Controls | Month 0
  mg/dL
Low-density lipoprotein in Controls | Month 3
  mg/dL
Low-density lipoprotein in Controls | Month 6
  mg/dL
High-density lipoprotein in the Experimental Group | Month 0
  mg/dL
High-density lipoprotein in the Experimental Group | Month 3
  mg/dL
High-density lipoprotein in the Experimental Group | Month 6
  mg/dL
High-density lipoprotein in Controls | Month 0
  mg/dL
High-density lipoprotein in Controls | Month 3
  mg/dL
High-density lipoprotein in Controls | Month 6
  mg/dL
Triglycerides in the Experimental Group | Month 0
  mg/dL
Triglycerides in the Experimental Group | Month 3
  mg/dL
Triglycerides in the Experimental Group | Month 6
  mg/dL
Triglycerides in Controls | Month 0
  mg/dL
Triglycerides in Controls | Month 3
  mg/dL
Triglycerides in Controls | Month 6
  mg/dL
Blood glucose levels in the Experimental Group | Month 0
  mg/dL
Blood glucose levels in the Experimental Group | Month 3
  mg/dL
Blood glucose levels in the Experimental Group | Month 6
  mg/dL
Blood glucose levels in Controls | Month 0
  mg/dL
Blood glucose levels in Controls | Month 3
  mg/dL
Blood glucose levels in Controls | Month 6
  mg/dL
Compliance with medication in the Experimental Group | Month 0
  YES/NO
Compliance with medication in the Experimental Group | Month 3
  YES/NO
Compliance with medication in the Experimental Group | Month 6
  YES/NO
Compliance with medication in Controls | Month 0
  YES/NO
Compliance with medication in Controls | Month 3
  YES/NO
Compliance with medication in Controls | Month 6
  YES/NO
Motivation for doing physical activity in the Experimental Group | Month 0
  The EMAPS scale (Echelle de Motivation envers l'Activité Physique en contexte de Santé = Scale for Motivation for Physical Activity in the Context of Health).This is an 18-item questionnaire with scores from 1 to 7. Depending on the patient's answers to the questions, the type and extent of motivation are defined. Score 18 - 126
Motivation for doing physical activity in the Experimental Group | Month 3
  The EMAPS scale (Echelle de Motivation envers l'Activité Physique en contexte de Santé = Scale for Motivation for Physical Activity in the Context of Health).This is an 18-item questionnaire with scores from 1 to 7. Depending on the patient's answers to the questions, the type and extent of motivation are defined. Score 18 - 126
Motivation for doing physical activity in the Experimental Group | Month 6
  The EMAPS scale (Echelle de Motivation envers l'Activité Physique en contexte de Santé = Scale for Motivation for Physical Activity in the Context of Health).This is an 18-item questionnaire with scores from 1 to 7. Depending on the patient's answers to the questions, the type and extent of motivation are defined. Score 18 - 126
Motivation for doing physical activity in Controls | Month 0
  The EMAPS scale (Echelle de Motivation envers l'Activité Physique en contexte de Santé = Scale for Motivation for Physical Activity in the Context of Health).This is an 18-item questionnaire with scores from 1 to 7. Depending on the patient's answers to the questions, the type and extent of motivation are defined. Score 18 - 126
Motivation for doing physical activity in Controls | Month 3
  The EMAPS scale (Echelle de Motivation envers l'Activité Physique en contexte de Santé = Scale for Motivation for Physical Activity in the Context of Health).This is an 18-item questionnaire with scores from 1 to 7. Depending on the patient's answers to the questions, the type and extent of motivation are defined. Score 18 - 126
Motivation for doing physical activity in Controls | Month 6
  The EMAPS scale (Echelle de Motivation envers l'Activité Physique en contexte de Santé = Scale for Motivation for Physical Activity in the Context of Health).This is an 18-item questionnaire with scores from 1 to 7. Depending on the patient's answers to the questions, the type and extent of motivation are defined. Score 18 - 126
Exercise Confidence Survey in the Experimental Group | Month 0
  French version of the "Exercise Confidence Survey" for regular physical activity) according to Eeckhout et al. 2012. The ECS questionnaire measures perceived self-efficacy for regular physical activity. It has two dimensions in the Exercise Confidence Survey: "sticking to it" and "making time for exercise". The survey has 8 questions to be answered by "I Know I can" (1 point) "Maybe I can" (3 points) or "I Know I cannot" (5 points). (Sallis et al., 1996)
Exercise Confidence Survey in the Experimental Group | Month 3
  French version of the "Exercise Confidence Survey" for regular physical activity) according to Eeckhout et al. 2012. The ECS questionnaire measures perceived self-efficacy for regular physical activity. It has two dimensions in the Exercise Confidence Survey: "sticking to it" and "making time for exercise". The survey has 8 questions to be answered by "I Know I can" (1 point) "Maybe I can" (3 points) or "I Know I cannot" (5 points). (Sallis et al., 1996)
Exercise Confidence Survey in the Experimental Group | Month 6
  French version of the "Exercise Confidence Survey" for regular physical activity) according to Eeckhout et al. 2012. The ECS questionnaire measures perceived self-efficacy for regular physical activity. It has two dimensions in the Exercise Confidence Survey: "sticking to it" and "making time for exercise". The survey has 8 questions to be answered by "I Know I can" (1 point) "Maybe I can" (3 points) or "I Know I cannot" (5 points). (Sallis et al., 1996)
Exercise Confidence Survey in Controls | Month 0
  French version of the "Exercise Confidence Survey" for regular physical activity) according to Eeckhout et al. 2012. The ECS questionnaire measures perceived self-efficacy for regular physical activity. It has two dimensions in the Exercise Confidence Survey: "sticking to it" and "making time for exercise". The survey has 8 questions to be answered by "I Know I can" (1 point) "Maybe I can" (3 points) or "I Know I cannot" (5 points). (Sallis et al., 1996)
Exercise Confidence Survey in Controls | Month 3
  French version of the "Exercise Confidence Survey" for regular physical activity) according to Eeckhout et al. 2012. The ECS questionnaire measures perceived self-efficacy for regular physical activity. It has two dimensions in the Exercise Confidence Survey: "sticking to it" and "making time for exercise". The survey has 8 questions to be answered by "I Know I can" (1 point) "Maybe I can" (3 points) or "I Know I cannot" (5 points). (Sallis et al., 1996)
Exercise Confidence Survey in Controls | Month 6
  French version of the "Exercise Confidence Survey" for regular physical activity) according to Eeckhout et al. 2012. The ECS questionnaire measures perceived self-efficacy for regular physical activity. It has two dimensions in the Exercise Confidence Survey: "sticking to it" and "making time for exercise". The survey has 8 questions to be answered by "I Know I can" (1 point) "Maybe I can" (3 points) or "I Know I cannot" (5 points). (Sallis et al., 1996)
Mediterranean diet adherence test in the Experimental Group | Month 0
  The MEDAS (Mediterranean diet Adherence Screener) score is a 14-point self-administered questionnaire used to assess adherence to a Mediterranean diet, based on consumption thresholds for 11 food groups (olive oil, vegetables, fruit, red meat, butter or cream, sweetened beverages, wine, legumes, fish, pastries and nuts), plus an additional question on preferential consumption of red or white meat. A score of 9 or over proves adherence to the Mediterranean diet.
Mediterranean diet adherence test in the Experimental Group | Month 3
  The MEDAS (Mediterranean diet Adherence Screener) score is a 14-point self-administered questionnaire used to assess adherence to a Mediterranean diet, based on consumption thresholds for 11 food groups (olive oil, vegetables, fruit, red meat, butter or cream, sweetened beverages, wine, legumes, fish, pastries and nuts), plus an additional question on preferential consumption of red or white meat. A score of 9 or over proves adherence to the Mediterranean diet.
Mediterranean diet adherence test in the Experimental Group | Month 6
  The MEDAS (Mediterranean diet Adherence Screener) score is a 14-point self-administered questionnaire used to assess adherence to a Mediterranean diet, based on consumption thresholds for 11 food groups (olive oil, vegetables, fruit, red meat, butter or cream, sweetened beverages, wine, legumes, fish, pastries and nuts), plus an additional question on preferential consumption of red or white meat. A score of 9 or over proves adherence to the Mediterranean diet.
Mediterranean diet adherence test in Controls | Month 0
  The MEDAS (Mediterranean diet Adherence Screener) score is a 14-point self-administered questionnaire used to assess adherence to a Mediterranean diet, based on consumption thresholds for 11 food groups (olive oil, vegetables, fruit, red meat, butter or cream, sweetened beverages, wine, legumes, fish, pastries and nuts), plus an additional question on preferential consumption of red or white meat. A score of 9 or over proves adherence to the Mediterranean diet.
Mediterranean diet adherence test in Controls | Month 3
  The MEDAS (Mediterranean diet Adherence Screener) score is a 14-point self-administered questionnaire used to assess adherence to a Mediterranean diet, based on consumption thresholds for 11 food groups (olive oil, vegetables, fruit, red meat, butter or cream, sweetened beverages, wine, legumes, fish, pastries and nuts), plus an additional question on preferential consumption of red or white meat. A score of 9 or over proves adherence to the Mediterranean diet.
Mediterranean diet adherence test in Controls | Month 6
  The MEDAS (Mediterranean diet Adherence Screener) score is a 14-point self-administered questionnaire used to assess adherence to a Mediterranean diet, based on consumption thresholds for 11 food groups (olive oil, vegetables, fruit, red meat, butter or cream, sweetened beverages, wine, legumes, fish, pastries and nuts), plus an additional question on preferential consumption of red or white meat. A score of 9 or over proves adherence to the Mediterranean diet.
Understanding barriers to motivation: Experimental group | Month 0
  The main barriers to physical activity cited by patients, and the responses provided by the healthcare professional - peer helper as part of therapeutic education sessions will be identified. Qualitative research
Understanding barriers to motivation: Experimental group | Month 3
  The main barriers to physical activity cited by patients, and the responses provided by the healthcare professional - peer helper as part of therapeutic education sessions will be identified. Qualitative research
Understanding barriers to motivation: Experimental group | Month 6
  The main barriers to physical activity cited by patients, and the responses provided by the healthcare professional - peer helper as part of therapeutic education sessions will be identified. Qualitative research
Understanding barriers to motivation in Controls | Month 0
  The main barriers to physical activity cited by patients, and the responses provided by the healthcare professional - peer helper as part of therapeutic education sessions will be identified. Qualitative research
Understanding barriers to motivation in Controls | Month 3
  The main barriers to physical activity cited by patients, and the responses provided by the healthcare professional - peer helper as part of therapeutic education sessions will be identified. Qualitative research
Understanding barriers to motivation in Controls | Month 6
  The main barriers to physical activity cited by patients, and the responses provided by the healthcare professional - peer helper as part of therapeutic education sessions will be identified. Qualitative research

CONTACTS AND LOCATIONS:
Overall Officials: Virginie VALLAYER, Principal Investigator — Nîmes University Hospital
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual-level data, including accelerometry recordings and questionnaire responses
Supporting Information: ICF
Time Frame: After completion of the primary analysis
Access Criteria: Upon reasonable request. Requests should be directed to the study's principal investigator and will require a data access agreement, in accordance with applicable ethical and data protection regulations

REFERENCES:
- [Background] Homs AF, Lachaux R, Vallayer V, Oulad Chrif K, Croizer M, Eglin I, Pionnier R, Chevallier T, Belvisi C, Dupeyron AF. Effects of a remote therapeutic education programme involving peers and health professionals on physical activity in patients with coronary heart disease undergoing phase 3 cardiac rehabilitation: protocol for a single-centre randomised controlled trial. BMJ Open. 2025 Jun 6;15(6):e095196. doi: 10.1136/bmjopen-2024-095196. PMID 40480674